CLINICAL TRIAL: NCT04822896
Title: Comparison of Acute Effects of Motor Imagery and Physical Exercise on Tongue Strength and Pain Threshold in Healthy Adults
Brief Title: Acute Effects of Motor Imagery and Physical Exercise on Tongue Strength and Pain Threshold in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5857-GOA
Record Dates: First submitted 2021-03-21; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Motor Imagery Training; Physical Exercise; Orofacial Exercise
Keywords: motor imagery; tongue strength; orofacial exercises
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesthetic Motor Imagery (Experimental): They will be asked to imagine the exercises kinesthetically from a first person perspective (as if they were doing it themselves).
  Interventions: Behavioral: Kinesthetic Motor Imagery Exercises
- Visual Motor Imagery (Experimental): They will be asked to imagine the exercises visually from a third person perspective (as if they were watching from the mirror / from the mirror while doing it themselves).
  Interventions: Behavioral: Visual Motor Imagery Exercises
- Real Physical Movements (Active Comparator): They will be asked to actually do the exercises shown in the video.
  Interventions: Behavioral: Physical Exercise

INTERVENTIONS:
Behavioral: Physical Exercise — The videos will be prepared by the researchers and will be watched by the physical exercise group, which includes exercises such as "shifting the jaw to the side, pushing the tongue forward, jaw opening, sliding the jaw with the tongue, opening the chin with the tongue, opening the chin by pressing the tongue against the palate and shifting the chin with the person's own resistance". Then they will be asked to do the exercises physically. Each exercise will be applied as 2 sets x 10 repetitions. There will be a 30-second break between sets.
  Arms: Real Physical Movements
Behavioral: Kinesthetic Motor Imagery Exercises — Seven exercises designated as "jaw shifting, tongue pushing forward, jaw opening, jaw shifting with tongue, jaw opening with tongue, jaw shifting by pressing the tongue on the palate, and chin shifting with one's own resistance", the videos prepared by the researchers and containing these exercises Once viewed, it will be applied as "kinesthetic imagery". Each exercise will be applied as 2 sets x 10 repetitions. There will be a 30-second break between sets.
  Arms: Kinesthetic Motor Imagery
Behavioral: Visual Motor Imagery Exercises — Seven exercises designated as "jaw shifting, tongue pushing forward, jaw opening, jaw shifting with tongue, jaw opening with tongue, jaw shifting by pressing the tongue on the palate, and chin shifting with one's own resistance", the videos prepared by the researchers and containing these exercises Once viewed, it will be applied as "visual imagery". Each exercise will be applied as 2 sets x 10 repetitions. There will be a 30-second break between sets.
  Arms: Visual Motor Imagery

SUMMARY:
Motor imagery is the feeling and thinking that the movement is done by imagination without physically occurring. In addition to its use in various fields, its use in the field of physiotherapy is also increasing. Especially in situations where real movement is difficult or contraindicated, motor visualization is very advantageous when there is no physical contact.

Swallowing function is one of the vital functions that ensure human independence. Like many components in swallowing, tongue muscle is also important. It has been shown that the strength of the tongue decreases with age, disease or other reasons. In the development of the strength of the tongue, while physiological principles are taken as basis, a different procedure from normal procedures is performed. However, language is a part of the body where one can study on his own.

Such situations lead to research on whether language reinforcement can occur with motor imagery. Considering that in addition to long-term effects, acute effects may also affect the functions of individuals, the starting point of the study is formed. Studies have investigated the acute change in tongue strength and pain perception after motor imagery.

The primary aim of this study is compare the acute effects of different motor imagery methods and physical exercise on tongue strength and pain in heatlhy adults.

ELIGIBILITY:
Inclusion Criteria:

* Participants age between 18-65
* Symmetrical chewing function, fluent mouth and tongue movements

Exclusion Criteria:

* Participants with systemic, cardiorespiratuar, central nerve system and romatologic diseases or musculoskeletal pain or craniocervical pathology
* A history of orofacial pain or temporomandibular diseases.
* Over-reacting for touching or tooth-pain
* Pregnancy or possibility of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in Tongue Strength | The outcome will be assessed at baseline and immediately after intervention.
  Tongue strength will be measured by the tongue pressure measuring device. The measurement will be in the form of placing a bulb filled with air and designed to transmit pressure, just behind the anterior teeth, on the hard palate, and the tongue compresses this bulb and transmits the pressure to the device. People will be asked to lift their tongue and press the bulbous for about three seconds. 3 measurements will be made in front and back of the tongue separately. In the anterior tongue evaluation, the bulb is placed in the palate just behind the teeth, and in the posterior tongue evaluation, the bulb is placed in the hard palate. It has been shown that it is valid and safe to measure the strength of the front and back regions of the tongue by this method.Measurements are recorded in kPa. The value of change in tongue strength expresses the effect of intervention on tongue strength. Higher kPa values mean strong tongue. Increasing in change implies that more force is being generated.
Change in Pain Threshold | The outcome will be assessed at baseline and immediately after intervention.
  Pain threshold will be measured with an algometer. The areas to be measured in this study were determined as masseter muscle (2.5 cm in front of the tragus, 1.5 cm below) and temporalis (3 cm above the lateral edge of the eye). Measurements from each region will be made 3 times at 30 second intervals and the average of the measurements will be included for analysis. During the measurement, the algometer will be held perpendicular to the skin. Measurement is terminated at the first value at which discomfort is felt. Measurements from each region will be made 3 times at 30 second intervals and the average of the measurements will be included for analysis. The change in pain threshold will be used as a measurement tool to determine how the intervention is affecting the pain threshold. Higher values in the pain threshold indicate that the person is more susceptible to pain.

SECONDARY OUTCOMES:
Change in Perceived Exertion | The outcome will be assessed at baseline and immediately after intervention.
  After the actual and motor imagery exercises, the perceived exertion of the participants will be evaluated with the Borg scale. On this scale, individuals rate their perceived difficulty between 6 (I did not feel any difficulty) and 20 (very, very difficult). High score means more perceived exertion.
Movement Imagery Questionnaire-Revised | At baseline
  It is a questionnaire used for administration in healthy adults and athletic populations and includes movements that require a high degree of skill and coordination. The visual and kinesthetic motor imagery skills of the person are measured with the scale consisting of 8 items. Items related to visual imagery are evaluated with a Likert type scale between 1 (very difficult to see) and 7 (very easy to see). Items related to kinesthetic imagery are likewise evaluated using a Likert-type scale that is graded between 1 (very difficult to feel) and 7 (very easy to feel). High scores indicate high visual and kinesthetic imagery skills. The Turkish validation study of the questionnaire has been conducted and it has been shown to be valid and reliable.
Mental Chronometer Time Ratio for Jaw Movement Task | At baseline
  The participants will actually execute and imagine a motor task: jaw movements. The duration of actual and imagined movements will be recorded by means of an electronic stopwatch. During the execution of the actual and imagined movements subjects will hold the electronic stopwatch in their non-dominant hand. They will start the stopwatch when they started to move (actual or imagined movement) and they will stop it when they completed their movement (actual or imagined). The ratio between real and imagined time will be calculated. A ratio close to 1 means that motor imagery is close to physical motion.
Mental Chronometer Time Ratio for Tongue Movement Task | At baseline
  The participants will actually execute and imagine a motor task: tongue movements. The duration of actual and imagined movements will be recorded by means of an electronic stopwatch. During the execution of the actual and imagined movements subjects will hold the electronic stopwatch in their non-dominant hand. They will start the stopwatch when they started to move (actual or imagined movement) and they will stop it when they completed their movement (actual or imagined). The ratio between real and imagined time will be calculated. A ratio close to 1 means that motor imagery is close to physical motion.
Mental Chronometer Time Ratio for Writing Task | At baseline
  The participants will actually execute and imagine a motor task: writing the following sentence: "Ankara is the capital of Turkey". The duration of actual and imagined movements will be recorded by means of an electronic stopwatch. During the execution of the actual and imagined movements subjects will hold the electronic stopwatch in their non-dominant hand. They will start the stopwatch when they started to move (actual or imagined movement) and they will stop it when they completed their movement (actual or imagined). A ratio close to 1 means that motor imagery is close to physical motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No